CLINICAL TRIAL: NCT03096184
Title: A Non-randomized Phase II Study of Apatinib Mesylate Tablets Plus Tegafur Gimeracil Oteracil Potassium Capsules in Recurrent/Metastatic Squamous Cell Carcinoma of Head and Neck
Brief Title: A Study of Apatinib Plus Tegafur Gimeracil Oteracil in Recurrent/Metastatic Head and Neck Cancers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Guopei Zhu, M.D., Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017HNRT001
Record Dates: First submitted 2017-03-25; First posted 2017-03-30 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: head and neck cancer; Apatinib; Tegafur Gimeracil Oteracil
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): Apatinib Mesylate Tablets and Tegafur Gimeracil Oteracil Potassium Capsules administered as a daily oral treatment
  Interventions: Drug: Apatinib Mesylate Tablets; Drug: Tegafur Gimeracil Oteracil Potassium Capsules

INTERVENTIONS:
Drug: Apatinib Mesylate Tablets — 500 mg qd.p.o. every day for 21 days as a cycle
  Other Names: Aitan
Drug: Tegafur Gimeracil Oteracil Potassium Capsules — 50mg bid p.o. every day for 14 days as a cycle
  Other Names: Aiyi

SUMMARY:
This is a non-randomized, phase II, open label study of apatinib mesylate tablets plus tegafur gimeracil oteracil potassium capsules in recurrent/metastatic squamous cell carcinoma of head and neck. The primary purpose of this study is to evaluate the efficacy of apatinib mesylate tablets plus tegafur gimeracil oteracil potassium capsules in recurrent/metastatic squamous cell carcinoma of head and neck

ELIGIBILITY:
Inclusion Criteria:

1. Histologically / cytologically confirmed diagnosis of recurrent or metastatic squamous cell carcinoma of head and neck origin not amenable to curative intent therapy; both human papillomavirus (HPV)(+) and HPV(-) tumors are eligible; tumors (squamous histology) of unknown primary that are clearly related to the head and neck area are eligible
2. Presence of measurable lesions (RECIST V1.1)
3. Eastern Cooperative Oncology Group (ECOG) performance status =< 2
4. Absolute neutrophil count (ANC) >= 1.5 x 10^9/L

   * Platelets >= 100 x 10^9/L
   * Hemoglobin (Hb) > 9 g/dL
   * Total calcium (corrected for serum albumin) within normal limits
   * Magnesium >= the lower limit of normal for the institution
   * Potassium within normal limits for the institution
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) within 1.5 x normal range (or =< 3.0 x upper limit of normal [ULN] if liver metastases are present)
   * Serum bilirubin within normal range (or =< 1.5 x ULN if liver metastases are present; or total bilirubin =< 3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert syndrome)
   * Serum creatinine =< 1.5 x ULN or 24-hour clearance >= 50 mL/min
   * Serum amylase =< ULN
   * Serum lipase =< ULN
   * Fasting plasma glucose =< 120 mg/dL (6.7 mmol/L)
5. Negative serum pregnancy test within 72 hours before starting study treatment in women with childbearing potential
6. Signed informed consent

Exclusion Criteria:

1. Patients with poor-controlled arterial hypertension (systolic pressure ≥ 140 mmHg and/or diastolic pressure ≥ 90 mm Hg) despite standard medical management;
2. Suffered from grade II or above myocardial ischemia or myocardial infarction, uncontrolled arrhythmias (including QT interval male ≥ 450 ms, female ≥ 470 ms). Grade III-IV cardiac insufficiency according to New York Heart Association (NYHA) criteria or echocardiography check: left ventricular ejection fraction (LVEF)<50%;
3. Patients who have had prior allergic reaction to Apatinib;
4. The subject has had another active malignancy within the past five years except for cervical cancer in site, in situ carcinoma of the bladder or non-melanoma carcinoma of the skin;
5. Clinically significant and uncontrolled major medical conditions including but not limited to: active uncontrolled infection, symptomatic congestive heart failure, Unstable angina pectoris or cardiac arrhythmia, psychiatric illness/ social situation that would limit compliance with study requirements; any medical condition, which in the opinion of the study investigator places the subject at an unacceptably high risk for toxicities;
6. Patients undergoing therapy with other investigational agents.
7. Women who are pregnant or breastfeeding;
8. Patients with any other concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2016-12-23 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | 2 years
  from date of enrollment until date of first documented disease progression or death from any cause, assessed up to 2 years
Overall survival | 2 years
  from date of enrollment until date of first death from any cause, assessed up to 2 years

SECONDARY OUTCOMES:
Acute toxicity profiles, graded according to the NCI CTCAE version 3.0 | 6 months
  Number of participants with treatment-related acute toxicity as assessed weekly by CTCAE v3.0 during the course of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai ninth people's hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No